CLINICAL TRIAL: NCT04776278
Title: Behavioral Economic and Wellness-based Approaches for Reducing Alcohol Use and Consequences Among Diverse Non-student Emerging Adults
Brief Title: Behavioral Economic and Wellness-based Approaches for Reducing Alcohol Use and Consequences Among Emerging Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Principal Investigator, James G Murphy, Professor, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AA029031 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-03-01 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Abuse
Keywords: Alcohol; Brief Intervention
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Methods; Relaxation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Brief Alcohol Intervention (BAI) + Substance Free Activity Session (SFAS) (Experimental): Participants first receive a 50-minute standard brief motivational intervention designed to reduce alcohol use. A week later, they will receive the Substance-free activity session (SFAS), a 50-minute counseling session designed to increase the salience of the individual's goals, to highlight the connection between their current patterns of behavior (including drinking and substance-free activities) and the attainment of these goals, and to increase future orientation and engagement in enjoyable and goal-directed activities that are inconsistent with substance use (even if the participant has no desire to change their use).
  Interventions: Behavioral: Brief Alcohol Intervention (BAI); Behavioral: Substance-free Activity Session (SFAS)
- Relaxation Training (RT) + Substance Free Activity Session (SFAS) (Experimental): Participants will complete a relaxation training session that will include a clinician leading them through a diaphragmatic breathing exercise, a progressive muscle relaxation protocol, and then a brief breath-counting (mindfulness) exercise. A week later, the participant will receive the SFAS, a 50-minute counseling session designed to increase the salience of the individual's goals, to highlight the connection between their current patterns of behavior (including drinking and substance-free activities) and the attainment of these goals, and to increase future orientation and engagement in enjoyable and goal-directed activities that are inconsistent with substance use (even if the participant has no desire to change their use).
  Interventions: Behavioral: Substance-free Activity Session (SFAS); Behavioral: Relaxation Training (RT)
- Education Control (Active Comparator): This minimal contact control condition will include a brief (2-3 minute) discussion where the research assistant (RA) who completed the assessment session will describe the educational handout. This condition is meant to approximate a public health-level approach to providing referral information and some of the content included in the BAI+SFAS condition but without any of the personalized information or motivational interviewing. Participants will receive information on risks associated with alcohol/drug misuse, strategies for reducing alcohol problems, managing stress, and goal-setting. The handout will also include links to hotlines, websites, and apps related to these domains. This condition will not include booster contact
  Interventions: Other: Education Control

INTERVENTIONS:
Behavioral: Brief Alcohol Intervention (BAI) — This session includes a discussion related to harm reduction and the participant's autonomy to make decisions about the information provided in the session; an alcohol use decisional balance exercise; personalized alcohol-related feedback, and goal-setting. Elements included in the feedback are: (a) comparison of the participant's perception of how much he or she drinks and actual norms, (b) a comparison of the participant's alcohol consumption vs. norms, (c) an estimate of the participant's peak blood alcohol content in the past month, (d) alcohol-related problems experienced, (e) money spent on alcohol, and (f) calories consumed from alcohol. Participants discuss the personalized feedback with the clinician and review protective behavioral strategies if he or she indicates interest.
  Arms: Brief Alcohol Intervention (BAI) + Substance Free Activity Session (SFAS)
Behavioral: Substance-free Activity Session (SFAS) — The SFAS session includes : a) discussion of life goals, b) discussion of associations between alcohol and drug use, goals, and substance-free activities; c) a graph depicting the participant's ratings of the relative importance of various aspects of their life and how their actions in the past week have been consistent with these priorities; d) personalized feedback on recent time allocation to activities across life domains, and a discussion of any changes the participant would like to make; e) feedback on symptoms of stress, anxiety and discussion of adaptive coping strategies; f) discussion of enjoyable substance-free activities and hobbies and substance-free recreational activity suggestions tailored to individual's interests and neighborhood; g) a goal setting exercise for specific behavior change plans; h) a Future Thinking Writing Exercise. Participants will receive weekly text-message based booster prompts for four weeks after their SFAS session.
  Arms: Brief Alcohol Intervention (BAI) + Substance Free Activity Session (SFAS); Relaxation Training (RT) + Substance Free Activity Session (SFAS)
Behavioral: Relaxation Training (RT) — The clinician will begin by establishing the credibility of the session by providing the participant with the rationale that developing relaxation or mindfulness training strategies can reduce stress and enhance wellness. The clinician will then lead the participant through a diaphragmatic breathing exercise, followed by a progressive muscle RT protocol, and then a brief breath-counting (mindfulness) exercise. The session will conclude with a brief discussion of additional stress and anxiety management strategies (e.g., apps to monitor heartrate and breathing). Participants will be asked about their reaction to the techniques and, if interested, encouraged to commit to a specific plan for practicing these techniques.
  Arms: Relaxation Training (RT) + Substance Free Activity Session (SFAS)
Other: Education Control — This condition will not include any clinical contact other than a brief (2-3 minute) discussion with the research assistant (RA) who completed the assessment session and who will describe the educational handout. This condition is meant to approximate a low-threshold public health-level approach to providing referral information and some of the content included in the BAI+SFAS condition but without any of the personalized information or MI/clinical contact. Thus, participants will receive information on risks associated with alcohol and drug misuse, strategies for reducing use/problems, and strategies for managing stress and setting and follow-through with achievable goals. The handout will also include links to hotlines, websites, and apps related to these domains. This condition will not include booster contact.
  Arms: Education Control

SUMMARY:
The purpose of this study is to evaluate an intervention approach for non-student emerging adults that attempts to reduce alcohol use by decreasing stress and increasing engagement in positive and goal-directed activities that provide meaningful alternatives to alcohol use.

DETAILED DESCRIPTION:
Brief alcohol interventions (BAI) are among the most cost-effective preventive care measures available and the evaluation of these interventions with high-risk and difficult-to-reach populations is an NIAAA priority. Although emerging adults (EAs) who attend college often have access to brief alcohol interventions (BAIs), there is a critical need to enhance both the efficacy and potential for dissemination of these approaches with high-risk non-student EAs. EAs who are not 4-year college students or graduates report higher levels of alcohol-related problems, greater levels of comorbid drug use and mental health symptoms, and higher risk for chronic alcohol use disorder compared to college graduates. Most BAIs include a single session focused explicitly on discussing risks associated with drinking and correcting normative beliefs about drinking rates without addressing the reasons why EAs may drink, including stress and limited behavioral alternatives to drinking. Because many EAs who do not graduate from college are socially and economically marginalized, an approach that encourages them to drink less without providing the tools to reduce stress and develop mood enhancing behavioral substitutes to drinking or drug use is unlikely to be successful. The Substance-Free Activity Session (SFAS) attempts to increase engagement goal-directed activities that might provide alternatives to alcohol use and also includes strategies for coping with stress/depression. The two-session (plus booster) BAI+SFAS approach has demonstrated efficacy for reducing both alcohol use/problems and depressive symptoms in two randomized clinical trials with college EAs and may be a more promising approach than single-session BAIs for higher-risk non-student EAs. Two critical next steps are to: 1) evaluate the BAI+SFAS with non-student EAs, and 2) determine if a two-session Relaxation Training (RT) +SFAS approach, which would enhance wellness and address two synergistic risk factors for alcohol misuse, demonstrates similar efficacy as the BAI+SFAS intervention. If so, this wellness-based approach may have greater potential for dissemination than approaches that include a BAI because the session content may be more appealing to EAs (managing stress and increasing positive activities). Thus, the primary goal of the proposed study is to establish the efficacy of these novel BAI approaches with high-risk community dwelling EAs, and a secondary goal is to identify factors that may increase potential for dissemination. We will conduct a randomized 3-group (BAI+SFAS vs. RT+SFAS vs. education control) trial with 525 EAs (175 per group; estimated 50% women & 50% African American) who report recent heavy drinking and who are not students or graduates of 4-year colleges. Outcomes will be assessed at 1, 3, 6, and 12 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 29 years old
* Not a current student or graduate of a 4-year college with no plans to enroll in a 4-year college in the upcoming semester
* Stable domicile and contact information
* Fluent English speaker
* Adequate literacy (>9th grade reading ability)
* Two or more heavy episodic drinking episodes in the past month (>5/4 standard drinks for males/ females) or exceeding NIAAA guidelines for high risk drinking (>14/7 drinks per week for men/women).

Exclusion Criteria:

* Current/past psychosis
* Current self-initiated AUD/SUD treatment
* Weekly or greater nonmedical use of prescription drugs or illegal drugs except cannabis
* Risk for alcohol withdrawal as evidenced by either 1) a recent history of alcohol withdrawal symptoms (tremors, anxiety, hallucinations, and seizures that occur after stopping drinking) or 2) very heavy weekly drinking reports on the alcohol screener (> 40 standard drinks in a typical week in the past month, a value that is > 2 standard deviations above the average drinks per week level observed in our previous brief alcohol intervention studies).

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 525 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Alcohol Consumption and Drug Use at 1-month | Enrollment, 1-month post intervention
  At each assessment point, participants will complete a computer administered Daily Drinking Questionnaire (DDQ) concerning their daily drinking during a typical week in the past month, an interval found sufficiently long to characterize drinking patterns.
Change from Baseline Alcohol Consumption and Drug Use at 3-months | Enrollment, 3-months post intervention
  At each assessment point, participants will complete a computer administered Daily Drinking Questionnaire (DDQ) concerning their daily drinking during a typical week in the past month, an interval found sufficiently long to characterize drinking patterns.
Change from Baseline Alcohol Consumption and Drug Use at 6-months | Enrollment, 6-months post-intervention
  At each assessment point, participants will complete a computer administered Daily Drinking Questionnaire (DDQ) concerning their daily drinking during a typical week in the past month, an interval found sufficiently long to characterize drinking patterns.
Change from Baseline Alcohol Consumption and Drug Use at 12-months | Enrollment, 12-months post intervention
  At each assessment point, participants will complete a computer administered Daily Drinking Questionnaire (DDQ) concerning their daily drinking during a typical week in the past month, an interval found sufficiently long to characterize drinking patterns.
Change from Baseline Alcohol-related Consequences at 1-month | Enrollment, 1-month
  The Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ) questionnaire asks about negative events over the past month (e.g., neglected obligations, driving after drinking). Research has shown that the BYAACQ is reliable yet sensitive to changes in alcohol use, has high internal consistency, and includes common but less severe consequences.
Change from Baseline Alcohol-related Consequences at 3-months | Enrollment, 3-months
  The Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ) questionnaire asks about negative events over the past month (e.g., neglected obligations, driving after drinking). Research has shown that the BYAACQ is reliable yet sensitive to changes in alcohol use, has high internal consistency, and includes common but less severe consequences.
Change from Baseline Alcohol-related Consequences at 6-months | Enrollment, 6-months
  The Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ) questionnaire asks about negative events over the past month (e.g., neglected obligations, driving after drinking). Research has shown that the BYAACQ is reliable yet sensitive to changes in alcohol use, has high internal consistency, and includes common but less severe consequences.
Change from Baseline Alcohol-related Consequences at 12-months | Enrollment, 12-months
  The Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ) questionnaire asks about negative events over the past month (e.g., neglected obligations, driving after drinking). Research has shown that the BYAACQ is reliable yet sensitive to changes in alcohol use, has high internal consistency, and includes common but less severe consequences.

SECONDARY OUTCOMES:
Change from Baseline Substance-free and Substance-related Activity Participation at 1-month | Enrollment, 1-month post intervention
  Participants report past month frequency and rate the enjoyment of 16 activities that are substance free vs. substance involved. Frequency and enjoyment ratings are multiplied to obtain a cross product that reflects reinforcement derived from the activity, and the relative reinforcement value of alcohol (R-ratio) is computed for analysis [(alcohol-related total / (alcohol-free total + alcohol-related total)]. Participants also report the number of hours spent engaging in several activity categories during a typical week in the past month (work, exercise, drinking, recreation). This information is used to generate the initial SFAS feedback on time allocation and potential alternatives to drinking and, at follow-up, will evaluate whether the interventions resulted in increased participation in substance-free activities, increased substance-free reinforcement, and decreased proportionate substance-related reinforcement relative to the control condition (R-ratio).
Change from Baseline Substance-free and Substance-related Activity Participation at 3-months | Enrollment, 3-months post intervention
  Participants report past month frequency and rate the enjoyment of 16 activities that are substance free vs. substance involved. Frequency and enjoyment ratings are multiplied to obtain a cross product that reflects reinforcement derived from the activity, and the relative reinforcement value of alcohol (R-ratio) is computed for analysis [(alcohol-related total / (alcohol-free total + alcohol-related total)]. Participants also report the number of hours spent engaging in several activity categories during a typical week in the past month (work, exercise, drinking, recreation). This information is used to generate the initial SFAS feedback on time allocation and potential alternatives to drinking and, at follow-up, will evaluate whether the interventions resulted in increased participation in substance-free activities, increased substance-free reinforcement, and decreased proportionate substance-related reinforcement relative to the control condition (R-ratio).
Change from Baseline Substance-free and Substance-related Activity Participation at 6-months | Enrollment, 6-months post intervention
  Participants report past month frequency and rate the enjoyment of 36 activities that are substance free vs. substance involved. Frequency and enjoyment ratings are multiplied to obtain a cross product that reflects reinforcement derived from the activity, and the relative reinforcement value of alcohol (R-ratio) is computed for analysis [(alcohol-related total / (alcohol-free total + alcohol-related total)]. Participants also report the number of hours spent engaging in several activity categories during a typical week in the past month (work, exercise, drinking, recreation). This information is used to generate the initial SFAS feedback on time allocation and potential alternatives to drinking and, at follow-up, will evaluate whether the interventions resulted in increased participation in substance-free activities, increased substance-free reinforcement, and decreased proportionate substance-related reinforcement relative to the control condition (R-ratio).
Change from Baseline Substance-free and Substance-related Activity Participation at 12-months | Enrollment, 12-months post intervention
  Participants report past month frequency and rate the enjoyment of 16 activities that are substance free vs. substance involved. Frequency and enjoyment ratings are multiplied to obtain a cross product that reflects reinforcement derived from the activity, and the relative reinforcement value of alcohol (R-ratio) is computed for analysis [(alcohol-related total / (alcohol-free total + alcohol-related total)]. Participants also report the number of hours spent engaging in several activity categories during a typical week in the past month (work, exercise, drinking, recreation). This information is used to generate the initial SFAS feedback on time allocation and potential alternatives to drinking and, at follow-up, will evaluate whether the interventions resulted in increased participation in substance-free activities, increased substance-free reinforcement, and decreased proportionate substance-related reinforcement relative to the control condition (R-ratio).
Change from Baseline Alcohol Purchase Task responses at 1-month | Enrollment, 1-month post intervention
  This questionnaire asks participants to report how many standard drinks they would consume across 20 prices ($0 to $20) in an imaginary drinking setting, which yields multiple observed and derived indices reflecting sensitivity to price changes that correspond with actual alcohol use. Elasticity of demand and intensity (consumption at $0) will be used for analysis. Relative insensitivity to price changes ("inelastic" demand) is related to risky drinking and alcohol problems, and intensity has incremental utility to predict alcohol use disorder symptoms beyond drinking practices. Consistent with previous research, alcohol demand will be evaluated as a mediator of treatment outcomes.
Change from Baseline Alcohol Purchase Task responses at 3-months | Enrollment, 3-months post intervention
  This questionnaire asks participants to report how many standard drinks they would consume across 20 prices ($0 to $20) in an imaginary drinking setting, which yields multiple observed and derived indices reflecting sensitivity to price changes that correspond with actual alcohol use. Elasticity of demand and intensity (consumption at $0) will be used for analysis. Relative insensitivity to price changes ("inelastic" demand) is related to risky drinking and alcohol problems, and intensity has incremental utility to predict alcohol use disorder symptoms beyond drinking practices. Consistent with previous research, alcohol demand will be evaluated as a mediator of treatment outcomes.
Change from Baseline Alcohol Purchase Task responses at 6-months | Enrollment, 6-months post intervention
  This questionnaire asks participants to report how many standard drinks they would consume across 20 prices ($0 to $20) in an imaginary drinking setting, which yields multiple observed and derived indices reflecting sensitivity to price changes that correspond with actual alcohol use. Elasticity of demand and intensity (consumption at $0) will be used for analysis. Relative insensitivity to price changes ("inelastic" demand) is related to risky drinking and alcohol problems, and intensity has incremental utility to predict alcohol use disorder symptoms beyond drinking practices. Consistent with previous research, alcohol demand will be evaluated as a mediator of treatment outcomes.
Change from Baseline Alcohol Purchase Task responses at 12-months | Enrollment, 12-months post intervention
  This questionnaire asks participants to report how many standard drinks they would consume across 20 prices ($0 to $20) in an imaginary drinking setting, which yields multiple observed and derived indices reflecting sensitivity to price changes that correspond with actual alcohol use. Elasticity of demand and intensity (consumption at $0) will be used for analysis. Relative insensitivity to price changes ("inelastic" demand) is related to risky drinking and alcohol problems, and intensity has incremental utility to predict alcohol use disorder symptoms beyond drinking practices. Consistent with previous research, alcohol demand will be evaluated as a mediator of treatment outcomes.
Change from Baseline in the Depression, Anxiety, and Stress Scales (DASS) at 1-month | Enrollment, 1-month post intervention
  The DASS is a reliable and valid self-report survey designed to measure symptoms of depression, anxiety and stress. Each of the three DASS scales contains seven items and participants are asked to use 4-point scales to rate the extent to which they have experienced each emotional state over the past week; scores for depression, anxiety and stress are calculated by summing the scores. For the purpose of this study, we will only include the depression and anxiety subscale items. Previous research indicates that the BAI+SFAS is associated with decreases in DASS scores, and we will evaluate DASS subscale scores as a secondary outcome and mediator of treatment effects.
Change from Baseline in the Depression, Anxiety, and Stress Scales (DASS) at 3-month | Enrollment, 3-months post intervention
  The DASS is a reliable and valid self-report survey designed to measure symptoms of depression, anxiety and stress. Each of the three DASS scales contains seven items and participants are asked to use 4-point scales to rate the extent to which they have experienced each emotional state over the past week; scores for depression, anxiety and stress are calculated by summing the scores. For the purpose of this study, we will only include the depression and anxiety subscale items. Previous research indicates that the BAI+SFAS is associated with decreases in DASS scores, and we will evaluate DASS subscale scores as a secondary outcome and mediator of treatment effects.
Change from Baseline in the Depression, Anxiety, and Stress Scales (DASS) at 6-months | Enrollment, 6-months post intervention
  The DASS is a reliable and valid self-report survey designed to measure symptoms of depression, anxiety and stress. Each of the three DASS scales contains seven items and participants are asked to use 4-point scales to rate the extent to which they have experienced each emotional state over the past week; scores for depression, anxiety and stress are calculated by summing the scores. For the purpose of this study, we will only include the depression and anxiety subscale items. Previous research indicates that the BAI+SFAS is associated with decreases in DASS scores, and we will evaluate DASS subscale scores as a secondary outcome and mediator of treatment effects.
Anxiety, and Stress Scales (DASS) at 12-months | Enrollment, 12-months post intervention
  The DASS is a reliable and valid self-report survey designed to measure symptoms of depression, anxiety and stress. Each of the three DASS scales contains seven items and participants are asked to use 4-point scales to rate the extent to which they have experienced each emotional state over the past week; scores for depression, anxiety and stress are calculated by summing the scores. For the purpose of this study, we will only include the depression and anxiety subscale items. Previous research indicates that the BAI+SFAS is associated with decreases in DASS scores, and we will evaluate DASS subscale scores as a secondary outcome and mediator of treatment effects.
Change from Baseline in the Short Self-Regulation Questionnaire (SSRQ) at 1-month | Enrollment, 1-month post intervention
  The SSRQ is a reliable and valid measure of the extent to which individuals are able to organize their behavior around the pursuit of goals and has been shown to mediate the drinking reductions associated with the SFAS. We will examine the SSRQ as a secondary intervention outcome and mediator.
Change from Baseline in the Short Self-Regulation Questionnaire (SSRQ) at 3-months | Enrollment, 3-months post intervention
  The SSRQ is a reliable and valid measure of the extent to which individuals are able to organize their behavior around the pursuit of goals and has been shown to mediate the drinking reductions associated with the SFAS. We will examine the SSRQ as a secondary intervention outcome and mediator.
Change from Baseline in the Short Self-Regulation Questionnaire (SSRQ) at 6-months | Enrollment, 6-months post intervention
  The SSRQ is a reliable and valid measure of the extent to which individuals are able to organize their behavior around the pursuit of goals and has been shown to mediate the drinking reductions associated with the SFAS. We will examine the SSRQ as a secondary intervention outcome and mediator.
Change from Baseline in the Short Self-Regulation Questionnaire (SSRQ) at 12-months | Enrollment, 12-months post intervention
  The SSRQ is a reliable and valid measure of the extent to which individuals are able to organize their behavior around the pursuit of goals and has been shown to mediate the drinking reductions associated with the SFAS. We will examine the SSRQ as a secondary intervention outcome and mediator.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Memphis, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will submit and share data with NIAAA Data Archive (NIAAADA), a data repository housed within the NIMH Data Archive (NDA). We also plan to release the data to qualified researchers who wish to collaborate with the study investigators. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: In this clinical trial, clinical assessments to establish baseline subject characteristics and eligibility criteria will be collected from all research participants at the screening and randomization visits, prior to the completion of the behavioral intervention. Assessment to measure changes in drinking and other dependent variables will take place a 1, 3, 6, and 12 months post-intervention.
Access Criteria: Qualified researchers

REFERENCES:
- [Derived] Murphy JG, Dennhardt AA, Tempchin J, Colgonis HE, McDevitt-Murphy ME, Borsari B, Berlin KS. Behavioral economic and wellness-based approaches for reducing alcohol use and consequences among diverse non-student emerging adults: study protocol for Project BLUE, a randomized controlled trial. Trials. 2024 Mar 9;25(1):173. doi: 10.1186/s13063-024-08009-9. PMID 38459579
- [Derived] Murphy JG, Dennhardt AA, Tempchin J, Colgonis HE, McDevitt-Murphy M, Borsari B, Berlin KS. Behavioral Economic and Wellness-based Approaches for Reducing Alcohol Use and Consequences Among Diverse Non-Student Emerging Adults: Study Protocol for Project BLUE, a Randomized Controlled Trial. Res Sq [Preprint]. 2024 Feb 7:rs.3.rs-3732598. doi: 10.21203/rs.3.rs-3732598/v1. PMID 38405755